CLINICAL TRIAL: NCT00209872
Title: Optimal Multimodal Analgesia in Abdominal Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMA-AH01; eudraCT # 2005-003595-38
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2005-09

CONDITIONS: Planned Abdominal Hysterectomy
MeSH Terms: interventions — Gabapentin; Lidocaine; Esketamine; Analgesia, Epidural

INTERVENTIONS:
Drug: Gabapentin
Drug: Lidocaine
Drug: S-ketamine
Procedure: Epidural analgesia

SUMMARY:
The purpose of this study is to test the current standard of care (SOC) treatment for abdominal hysterectomy with a group receiving SOC minus epidural analgesia plus additional perioperative analgesics in terms of postoperative abilities, postoperative nausea and vomiting (PONV), pain and discharge time from the PACU (post-anaesthesia care unit).

DETAILED DESCRIPTION:
Aim of the study: to compare postoperative complaints (PONV, pain, etc) and PACU discharge time between two groups, for patients admitted for planned abdominal hysterectomy with or without BSO:

* A: standard of care (SOC) receiving paracetamol, celecoxib, epidural analgesia, dexamethasone, ondansetron and droperidol, and general anaesthesia with propofol, remifentanil and cisatracurium
* B: SOC with sham epidural analgesia, preoperative gabapentin, intraoperative lidocaine, s-ketamine and sufentanil

ELIGIBILITY:
Inclusion Criteria:

* Planned abdominal hysterectomy with or without BSO
* Age above 18 years
* Written informed consent
* American Society of Anesthesiologists (ASA) class I-III

Exclusion Criteria:

* Planned vaginal or laparoscopic hysterectomy
* Hysterectomy as part of other surgery
* Allergy to part of the treatment regimen
* Previous reactions to opioids (nausea, cognition)
* Previous inability to place correct epidural catheter
* Severe state anxiety according to the OCAP or STAI
* ASA class IV
* Dependency on alcohol, opioids or central stimulants
* Chronic pain condition
* Hemorrhagic diathesis
* Participation in another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Postoperative abilities over time
Discharge time from PACU according to fixed criteria
Consumption of analgesics and antiemetics in the PACU

SECONDARY OUTCOMES:
Degree of nursing requirements at the PACU
General tolerability of the regimes
Threshold for sensory perception and pain using the Pain Matcher device, pre- and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, M.D., Principal Investigator — Dept. of Anaesthesia, Acute Pain Service, Hvidovre Hospital, Copenhagen, Denmark; Claus Lund, Dr. Med. Sci., Study Chair — Dept. of Anaesthesia, Hvidovre Hospital, Copenhagen, Denmark
Locations (1):
- Dept. of Anaesthesia, Hvidovre Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- See also: URL looking into anaesthesia and surgery for abdominal hysterectomy — http://www.postoppain.org